CLINICAL TRIAL: NCT01382979
Title: Evaluation of AlcoholEdu: A Randomized Multi-Campus Trial
Brief Title: Evaluation of AlcoholEdu for College
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Responsible Party: Mallie J. Paschall, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AA016584 (NIH)
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Alcohol Misuse
Keywords: Alcohol misuse prevention; College students; Intervention and control

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol education and prevention (Experimental): AlcoholEdu is an online course designed to prevent alcohol misuse and related problems among college freshmen.
  Interventions: Behavioral: AlcoholEdu for College
- Control (No Intervention): Control group.

INTERVENTIONS:
Behavioral: AlcoholEdu for College — Online course for college freshmen.
  Arms: Alcohol education and prevention

SUMMARY:
The study examined whether an online course for college freshmen (AlcoholEdu) had an effect on alcohol misuse and related problems, using a randomized controlled design with 30 universities.

ELIGIBILITY:
Inclusion Criteria:

* Colleges without an online alcohol prevention course
* Able to implement AlcoholEdu course for all incoming freshmen
* Able to provide random student samples for data collection
* Able to obtain IRB approval for study

Exclusion Criteria:

* Already implementing alcohol prevention course for incoming freshmen
* Not able to implement online alcohol prevention course
* Not able to provide random student samples for data collection
* Not able to obtain IRB approval for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9571 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Binge drinking | 30 days
  Frequency of binge drinking in the past 30 days

SECONDARY OUTCOMES:
Alcohol-related problems | 30 days
  Alcohol-related problems in the past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mallie J. Paschall, Ph.D., Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- Prevention Research Center, Berkeley, California, United States

REFERENCES:
- [Derived] Paschall MJ, Antin T, Ringwalt CL, Saltz RF. Evaluation of an Internet-based alcohol misuse prevention course for college freshmen: findings of a randomized multi-campus trial. Am J Prev Med. 2011 Sep;41(3):300-8. doi: 10.1016/j.amepre.2011.03.021. PMID 21855745